CLINICAL TRIAL: NCT06719596
Title: Probiotics Combined with Enteral Nutrition on Infectious Complications After Pancreaticoduodenectomy:a Single-centre, Prospective Randomised, Open, Parallel-controlled, Superiority Study
Brief Title: Probiotics Combined with Enteral Nutrition Reduces Postoperative Infectious Complications in PD
Acronym: 2024-225-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2024-225-01
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Infectious Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics combined with enteral nutrition reduces postoperative infectious complications in PD (Experimental): enteral nutrition+Pre-operative + one week post-operative Oral Bifidobacterium bifidum live triple capsule, 4 capsules Oral BID
  Interventions: Drug: Bifidobacterium Bifidum Oral Capsule
- Control group (No Intervention): Conventional postoperative treatment of the pancreas combined with enteral nutrition

INTERVENTIONS:
Drug: Bifidobacterium Bifidum Oral Capsule — enteral nutrition+Pre-operative + one week post-operative Oral Bifidobacterium bifidum live triple capsule, 4 capsules Oral BID
  Arms: Probiotics combined with enteral nutrition reduces postoperative infectious complications in PD

SUMMARY:
Probiotics combined with enteral nutrition reduces postoperative infectious complications in PD

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than 18 years of age;
* Indication for elective pancreaticoduodenal surgery;
* Patients who understand the nature of the trial and are willing and able to provide written consent

Exclusion Criteria:

. Current or recent (within the previous 1 month) use of probiotic-based products or antibiotic therapy medications.

Inability to tolerate PD due to cardiopulmonary function and other parameters

* Received radiotherapy before surgery
* Emergency PD surgery
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
infectious complication | 30 days after surgery
  1. Post-operative infections: Surgical site infections (SSI): including surgical incision infections and abdominal cavity infections.
  (1) incision infection: purulent secretions in the incision and culture of pathogenic bacteria (2) abdominal cavity infection: diagnosis can be made by meeting one of the following criteria: ① postoperative symptoms of systemic infection (fever > 38 ° C, white blood cell count higher than the upper limit of normal values), accompanied by abdominal distension, abdominal pain, and signs of peritonitis; ② abdominal drainage or puncture drainage fluid is purulent fluid, positive bacteriological culture results; ③ ultrasound, CT and other imaging tests or re-operation to confirm the presence of oozing or encapsulated abscess in the abdominal cavity; ③ ultrasound, CT and other imaging tests or re-operation to confirm the presence of oozing or encapsulated abscess. (iii) ultrasound or CT imaging or re-surgical confirmation of the presence of intra-abdominal ex

CONTACTS AND LOCATIONS:
Locations (1):
- 321 Zhongshan Road, Nanjing Gulou Hospital, Gulou District, Nanjing, Jiangsu Province, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided